CLINICAL TRIAL: NCT01066377
Title: A Randomised, Controlled, Parallel Study to Determine the Immunomodulatory Effects of Pre- and Probiotics Upon the Immune Response to Influenza Vaccination in Young and Older Volunteers
Brief Title: PRIMAGE (Probiotics, Immunity and Ageing)
Acronym: PRIMAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Reading (Other)
Responsible Party: Dr Mike Proven, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BB/H00470X/1
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: prebiotic; probiotic; influenza; vaccination; ageing; immunosenescence
MeSH Terms: conditions — Influenza, Human | interventions — Prebiotics; oligofructose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prebiotic and probiotic mix (Experimental): Prebiotic: 8g/day, will be selected on the basis of ability to promote optimal growth and survival of the probiotic (inulin, fructooligosaccharides [FOS], galactooligosaccharides[GOS] and xylooligosaccharides[XOS] will be tested). Probiotic: 10^8 - 10^9 live bacteria/day, bifidobacterium longum bv. infantis CCUG52486.
  Interventions: Dietary Supplement: Prebiotic and probiotic mix
- Maltodextrin/milk powder (Placebo Comparator)
  Interventions: Dietary Supplement: Prebiotic and probiotic mix

INTERVENTIONS:
Dietary Supplement: Prebiotic and probiotic mix — The probiotic strain will be Bifidobacterium longum bv. infantis CCUG 52486 (10^8 - 10^9 live bacteria per day), which was originally isolated from healthy elderly subjects, and which has been demonstrated to have particular ecological fitness and anti-pathogenic effects in vitro. A suitable prebiotic (8g/day) will be selected on the basis of ability to promote optimal growth and survival of this probiotic (inulin, fructooligosaccharides [FOS], galactooligosaccharides[GOS] and xylooligosaccharides[XOS] will be tested).
  Other Names: Bifidobacterium lactentis; Bifidobacterium liberorum; Bifidobacterium infantis; Bifidobacterium longum infantis; Bifidobacterium longum subsp. infantis; oligofructose; oligofructan; oligogalactosyllactose; oligogalactose; oligolactose; transgalactooligosacchariden

SUMMARY:
Ageing dramatically affects immune function; this phenomenon is known as immunosenescence and partly explains the increased susceptibility for infection in older individuals. Vaccination is recommended to protect older people against influenza, but immunosenescence also reduces the efficacy of vaccination. Probiotics are beneficial bacteria, which can be consumed and which have a long and safe record of use in humans. Often they are taken together with prebiotics, which are carbohydrates that provide a food source for the beneficial bacteria when they reach the lower gut. There is particular interest in the positive influences of pre- and probiotics in older people, who are subject to alteration in gut microflora composition as well as immunosenescence.

The PRIMAGE (Probiotics, immunity and ageing) study will examine the effect of a prebiotic and probiotic mix on the immune response to influenza vaccination in young and older subjects, and is funded by BBSRC DRINC. It will involve 60 young (18-35y) and 60 older (65-85y) subjects recruited from the local Reading community. Participants will take a pre- and probiotic mixture or a placebo for a total of 8 weeks. The probiotic is not currently commercially produced, but has been demonstrated to have particular ecological fitness and anti-pathogenic effects in the gastrointestinal tract in old age. A suitable prebiotic will be selected on the basis of ability to promote optimal growth and survival of this probiotic. After 4 weeks on the treatment, the subjects will receive an influenza vaccination. Blood, saliva and stool samples will be taken before treatment, and at 4, 6 and 8 weeks after commencement. The samples taken at 6 and 8 weeks will be used to assess the immune response to the vaccination. A wide range of immune parameters will be assessed, taking into account the age-related shifts in immune cell populations.

DETAILED DESCRIPTION:
The number of people aged 65 years and over is expected to rise by over 60% in the next 25 years, which presents an enormous challenge for the healthcare system. Ageing dramatically affects immune function; this phenomenon is known as immunosenescence and partly explains the increased susceptibility for infection in older individuals. Influenza is particularly common in older individuals and is a major cause of death in older people. Vaccination is recommended to protect elderly people against influenza, but immunosenescence also reduces the efficacy of vaccination. It has been estimated that 3050% of older adults fail to mount protective antibody responses after influenza vaccination, representing a considerable waste of resource and a false sense of security for those receiving the vaccinations.

Probiotics have shown promise in the prevention or treatment of several disease states ranging from lactose intolerance, constipation and diarrhoea, alleviation of allergy and even to more chronic systemic diseases, such as cardiovascular disease and cancer. Often they are taken together with prebiotics, which are carbohydrates that provide a food source for the beneficial bacteria when they reach the lower gut. There is particular interest in the positive influences of pre- and probiotics in older people, who are subject to alteration in gut microflora composition as well as immunosenescence. Several studies have demonstrated beneficial effects of specific pre- and probiotics on immune function in older subjects. However, none of these studies have taken into account the agerelated shift in immune cell populations. Furthermore, there is little understanding of the mechanisms underlying these effects. Despite this, probiotics have recently been proposed as prime candidates for 'antiimmunosenescence' therapy. We propose to investigate the impact of a pre- and probiotic mix on the immune response to influenza vaccination in young and older subjects, taking into account the age related shifts in immunity due to immunosenescence. The inclusion of both a young and older group of subjects will allow us to ascertain whether older individuals derive particular benefit from probiotics because of their altered gut microbiota and immune status.

This proposal brings together a unique combination of expertise in nutrition, gut health and immunology to determine the scientific basis for the immunomodulatory effects of pre- and probiotics. The chief investigator, Dr Parveen Yaqoob, has been working in the area of diet, health, ageing and immune function for 18 years. Professor Ian Rowland has been working on the interaction between diet and the gut microbiota and its implications for human health for 30 years. Dr Kieran Tuohy was appointed Lecturer in Food Metabonomics in the Department of Food Biosciences in 2005 and has over ten years experience in the field of gut microbiology and functional foods. Professor Margot Gosney is Director of Clinical Health Sciences, The University of Reading and a clinician working in elderly care at the Royal Berkshire NHS Foundation Trust, Reading. Her research interests include the association between nutrition and health of elderly people, ageing, oncology, dental science for stroke patients, influenza, incontinence, falls and intellectual decline. Dr Sue Todd is a Reader in Medical Statistics at the University of Reading and has over 15 years experience as an applied statistician working in the fields of clinical trials and epidemiology, with particular interest in sequential clinical trials, Data and Safety Monitoring Boards and statistical methods for epidemiology. Professor Richard Aspinall has been working on the hypothesis that age related changes in the T cell arm of the immune system are driven by age associated thymic atrophy. The Chief Investigator and the other project researchers have no direct personal involvement with the funding organisation (BBSRC DRINC) and therefore there are no conflicts of interest. The results of this study will also contribute to the PhD thesis of two postgraduate students.

Healthy volunteers (60 young [1835y] and 60 older [6585y]) will be randomly assigned to either a pre-and probiotic mix or to placebo (a maltodextrin/milk mix) for 8 weeks in total. The probiotic strain will be Bifidobacterium longum bv. infantis CCUG 52486 (10^8 10^9 live bacteria per day), which was originally isolated from healthy elderly subjects, and which has been demonstrated to have particular ecological fitness and antipathogenic effects in vitro. A suitable prebiotic (8g/day) will be selected on the basis of ability to promote optimal growth and survival of this probiotic (inulin, fructooligosaccharides [FOS], galactooligosaccharides[GOS] and xylooligosaccharides[XOS] will be tested). The pre- and probiotic mix and placebo sachet will be manufactured and packaged in the University of Reading pilot plant, and tested by Reading Scientific Services Limited for safety. This project will assess vaccine efficacy on the basis of both specific antibody titre and cellular responsiveness.

Participants will be required to visit the Department of Food and Nutritional Sciences on 5 occasions once for screening and 4 times during the study (0, 4, 6 and 8 weeks). The screening visit will involve a detailed medical history and several assessments to be conducted by a Research Nurse, making the visit approximately 2 hours duration. The study visits will be shorter (approximately 1 hour), involving a discussion of the study, identifying any problems or concerns and collection of biological samples. Blood (150ml), saliva and faecal samples will be collected at baseline and after 4 weeks of supplementation. After this sampling, subjects will receive an influenza vaccination (Solvay Pharmaceuticals) and further samples will be collected 2 and 4 weeks after vaccination.

ELIGIBILITY:
Inclusion Criteria:

Suitable study participants will be defined as:

* aged 18-35 (young cohort) or 65-85 (older cohort) men and women
* BMI 18.5 - 30 kg/m2
* good general health as determined by medical questionnaires and laboratory data from screening blood and urine sample (fasting glucose, ESR, FBC, liver function tests, renal profile, dipstick urinalysis)
* not pregnant, lactating or planning a pregnancy

Exclusion Criteria:

* allergy to the influenza vaccine
* HIV infection
* diabetes requiring any medication
* asplenia and other acquired or congenital immunodeficiencies
* any autoimmune disease
* malignancy
* cirrhosis
* connective tissue diseases
* current use of immunomodulating medication (including oral prednisone and inhaled steroids)
* self-reported symptoms of acute or recent infection (including use of antibiotics within last 3 months)
* taking lactulose or any other treatment for constipation
* alcoholism and drug misuse

Additional exclusion criteria for older volunteers includes:

* laboratory data which is outside the normal range for this age group AND outside the ranges specified in the SENIEUR protocol for ESR, FBC, renal profile, liver function tests, fasting glucose and dipstick urinalysis (Ligthart et al, 1984)
* Barthel Index score of <16
* CIRS score of <15.

Additional exclusion criteria for younger volunteers is:

* laboratory data which is outside the normal range
* influenza vaccination in the previous 12 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The immune response to influenza vaccination among young and older adults | 4 weeks after vaccination
  Serum vaccine-specific antibodies to the 2010-2011 influenza vaccine will be measured by hemagglutination assay.

SECONDARY OUTCOMES:
The cellular and molecular basis for modulation of immune function by pre- and probiotics. | Assessed after 4 weeks of pre- and probiotic treatment
  Blood samples will be subject to density gradient separation of peripheral blood mononuclear cells (PBMC), and cryopreserved for NK cell analysis, cell phenotypes, cytokine production, proliferation, expression of activation markers, expression of toll like receptors and assessment of T cell receptor excision circles (TREC). Serum and plasma will be stored for measurement of chemokines, plasma lipids and glucose. Saliva samples will be used to assess salivary IgA content.
The cellular and molecular basis for modulation of immune function by pre- and probiotics. | Assessed after 6 weeks of pre- and probiotic treatment
  Blood samples will be subject to density gradient separation of peripheral blood mononuclear cells (PBMC), and cryopreserved for NK cell analysis, cell phenotypes, cytokine production, proliferation, expression of activation markers, expression of toll like receptors and assessment of T cell receptor excision circles (TREC). Serum and plasma will be stored for measurement of chemokines, plasma lipids and glucose. Saliva samples will be used to assess salivary IgA content.
The cellular and molecular basis for modulation of immune function by pre- and probiotics. | Assessed after 8 weeks of pre- and probiotic treatment
  Blood samples will be subject to density gradient separation of peripheral blood mononuclear cells (PBMC), and cryopreserved for NK cell analysis, cell phenotypes, cytokine production, proliferation, expression of activation markers, expression of toll like receptors and assessment of T cell receptor excision circles (TREC). Serum and plasma will be stored for measurement of chemokines, plasma lipids and glucose. Saliva samples will be used to assess salivary IgA content.
The modulation of the gut microbiota by pre- and probiotics. | Assessed after 4 weeks of pre- and probiotic treatment
  Faecal samples will be processed for later analysis by fluorescence in situ hybridization (FISH) using oligonucleotide 16s rRNA probes targeting dominant and important groups of gut bacteria. Denatured gradient gel electrophoresis (DGGE) will be used to assess changes in faecal bacterial abundance and species diversity. qPCR will be used to identify specific bacterial species, including Bifidobacterium longum. Faecal dry weight and IgA content will be assessed. Faecal content of microbial metabolites such as short chain fatty acids and ammonia will be quantified.
The modulation of the gut microbiota by pre- and probiotics. | Assessed after 8 weeks of pre- and probiotic treatment
  Faecal samples will be processed for later analysis by fluorescence in situ hybridization (FISH) using oligonucleotide 16s rRNA probes targeting dominant and important groups of gut bacteria. Denatured gradient gel electrophoresis (DGGE) will be used to assess changes in faecal bacterial abundance and species diversity. qPCR will be used to identify specific bacterial species, including Bifidobacterium longum. Faecal dry weight and IgA content will be assessed. Faecal content of microbial metabolites such as short chain fatty acids and ammonia will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Parveen Yaqoob, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

REFERENCES:
- [Derived] Przemska-Kosicka A, Childs CE, Maidens C, Dong H, Todd S, Gosney MA, Tuohy KM, Yaqoob P. Age-Related Changes in the Natural Killer Cell Response to Seasonal Influenza Vaccination Are Not Influenced by a Synbiotic: a Randomised Controlled Trial. Front Immunol. 2018 Mar 22;9:591. doi: 10.3389/fimmu.2018.00591. eCollection 2018. PMID 29662493
- [Derived] Enani S, Przemska-Kosicka A, Childs CE, Maidens C, Dong H, Conterno L, Tuohy K, Todd S, Gosney M, Yaqoob P. Impact of ageing and a synbiotic on the immune response to seasonal influenza vaccination; a randomised controlled trial. Clin Nutr. 2018 Apr;37(2):443-451. doi: 10.1016/j.clnu.2017.01.011. Epub 2017 Jan 28. PMID 28215759
- [Derived] Przemska-Kosicka A, Childs CE, Enani S, Maidens C, Dong H, Dayel IB, Tuohy K, Todd S, Gosney MA, Yaqoob P. Effect of a synbiotic on the response to seasonal influenza vaccination is strongly influenced by degree of immunosenescence. Immun Ageing. 2016 Mar 15;13:6. doi: 10.1186/s12979-016-0061-4. eCollection 2016. PMID 26985232